CLINICAL TRIAL: NCT00001235
Title: Biochemical and Genetic Studies in Familial Alzheimer's Disease
Brief Title: Genetic Studies in Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 880029; 88-N-0029
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-02

CONDITIONS: Alzheimer's Disease; Nervous System Disease
Keywords: Primary Neuronal Degeneration; Genetics; Neurotransmitters; DNA; Lymphoblasts; Skin Fibroblast; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Nervous System Diseases

SUMMARY:
Alzheimer's disease is a condition marked by the deterioration of mental function. The disease usually begins in late middle life and results in death in 5 to 10 years. Patients with Alzheimer's disease typically suffer from memory loss, confusion, and disorientation. The condition has become a major medical and social problem in the United States because of the increasing number of people living beyond the age of 65. The actual cause of Alzheimer's disease is unknown.

Researchers believe that Alzheimer's disease, or at least a portion of cases, may be an inherited condition. As a result, many new techniques have been developed to study the genetic causes of Alzheimer's disease and other neurological disorders. Many of these genetic techniques require blood samples and a family pedigree. A pedigree is a chart, similar to a family tree, that shows a patient's family history.

The purpose of this study is to collect family and psychosocial information, blood, and biopsy samples from patients with neurological diseases, their families, and normal volunteers. This information gathered will be used to learn more about diseases that affect the brain.

DETAILED DESCRIPTION:
This is a screening and follow-up Protocol. Recent technological advances have facilitated the development of new approaches for investigating the underlying genetic basis of neurological disorders, but genetic questions remain open and on going. Application of many genetic techniques require a family pedigree and blood sample. Peripheral blood lymphoblasts which are banked also serve as a renewable source for harvesting DNA which can be used for developing genetic markers in the future. This study will allow collection of family and psychosocial information and blood specimens from patients with neurological diseases, their families, and normal control subjects.

ELIGIBILITY:
INCLUSION/EXCLUSION CRITERIA

Need to know extensive family history information.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Start 1988-02; Study Completion 2004-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Nee LE, Polinsky RJ, Eldridge R, Weingartner H, Smallberg S, Ebert M. A family with histologically confirmed Alzheimer's disease. Arch Neurol. 1983 Apr;40(4):203-8. doi: 10.1001/archneur.1983.04050040033004. PMID 6600923
- [Background] Sherrington R, Rogaev EI, Liang Y, Rogaeva EA, Levesque G, Ikeda M, Chi H, Lin C, Li G, Holman K, Tsuda T, Mar L, Foncin JF, Bruni AC, Montesi MP, Sorbi S, Rainero I, Pinessi L, Nee L, Chumakov I, Pollen D, Brookes A, Sanseau P, Polinsky RJ, Wasco W, Da Silva HA, Haines JL, Perkicak-Vance MA, Tanzi RE, Roses AD, Fraser PE, Rommens JM, St George-Hyslop PH. Cloning of a gene bearing missense mutations in early-onset familial Alzheimer's disease. Nature. 1995 Jun 29;375(6534):754-60. doi: 10.1038/375754a0. PMID 7596406
- [Background] Nee LE. Effects of psychosocial interactions at a cellular level. Soc Work. 1995 Mar;40(2):259-62. PMID 7732429